CLINICAL TRIAL: NCT01905384
Title: Randomized Controlled Trial Comparing Covered Versus Uncovered Metal Stents for Biliary Decompression in Inoperable Malignant Distal Bile Duct Obstruction
Brief Title: Covered vs Uncovered Metal Stents for Palliative Biliary Decompression in Inoperable Malignant Distal Bile Duct Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Patrick Yachimski, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 130331
Record Dates: First submitted 2013-05-29; First posted 2013-07-23 (Estimated); Results first posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Distal Bile Duct Obstruction
Keywords: pancreatic cancer; cholangiocarcinoma; metastatic malignancy; jaundice
MeSH Terms: conditions — Pancreatic Neoplasms; Cholangiocarcinoma; Neoplasms; Jaundice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- U-SEMS group (Active Comparator): Patients undergoing routine care ERCP and randomized to 10 mm diameter Uncovered Self-expanding metal biliary stents (U-SEMS) (Wallflex, Boston Scientific).
  Interventions: Device: Uncovered Self-expanding metal biliary stents (U-SEMS)
- C-SEMS Group (Active Comparator): Patients undergoing routine care ERCP and randomized to a 10 mm diameter Covered Self-Expanding metal biliary stents (C-SEMS) (Wallflex, Boston Scientific)
  Interventions: Device: Covered Self-expanding metal biliary stents (C-SEMS)

INTERVENTIONS:
Device: Covered Self-expanding metal biliary stents (C-SEMS) — Used for palliation of inoperable malignant distal bile duct obstruction.
  Arms: C-SEMS Group
Device: Uncovered Self-expanding metal biliary stents (U-SEMS) — Used for palliation of inoperable malignant distal bile duct obstructions.
  Arms: U-SEMS group

SUMMARY:
The purpose of this study is to compare the rate of long-term stent failure, defined as need for repeat biliary intervention following placement of C-SEMS vs U-SEMS for palliation of inoperable malignant distal bile duct obstruction.

ELIGIBILITY:
Inclusion Criteria:

* distal bile obstruction referred for ERCP with intended palliative metal stent placement for palliation of jaundice
* 18 years of age or older
* serum bilirubin > 2mg/dL

Exclusion Criteria:

* prior endoscopic or percutaneous biliary drainage
* post-surgical anatomy
* primary site of biliary obstruction involving the common hepatic duct or hilum
* tumor involving gastric outlet, duodenum, or ampulla either precluding endoscopic access to the papilla or otherwise preventing endoscopic biliary cannulation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Yachimski, MD, MPH, Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - Mount Sinai Hospital, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from patient population at the Vanderbilt Digestive Disease Center. Between November 8, 2017 until June 14, 2019, only 6 participants were randomized and completed the study.
Pre-assignment Details: 4 participants screen failed before being randomized to either arm of the study. Only 6 participants was randomized (3 to each arm) and completed the study.
Period: Overall Study
Arm/Group | U-SEMS Group | C-SEMS Group
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 3 participants were enrolled to each arm for a total of 6 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | U-SEMS Group | C-SEMS Group | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73 (0) | 73 (0) | 73 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 3 | 0 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Rate of Long-term Stent Failure
Description: Compare the rate of long-term stent failure, defined as need for repeat biliary intervention (endoscopic, percutaneous, or surgical) following placement of C-SEMS vs U-SEMS for palliation of inoperable malignant distal bile duct obstruction.
Time Frame: One year
Population: 3 participants randomized to each arm for a total of 6 participants. Of the 3 participants in the U-SEMS group, none needed repeat intervention. Of the 3 participants in the C-SEMS group, 2 needed repeat intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | U-SEMS Group | C-SEMS Group
Number analyzed (Participants) | 3 | 3
Participants | 0 | 2

2. Secondary Outcome: Rates of Adverse Stent-related or Intervention-related Outcomes
Description: Participants will be monitored for adverse stent-related or intervention-related outcomes such as pancreatitis, cholangitis, cholecystitis, perforation.
Time Frame: One Year
Population: 3 participants randomized to each arm for a total of 6 participants. Of the 3 participants in the U-SEMS group, there were no reports of pancreatitis, cholangitis, cholecystitis, or perforation. Of the 3 participants in the C-SEMS group, there were no reports of pancreatitis, cholangitis, cholecystitis, or perforation.
Measure: Count of Participants; unit: Participants
Arm/Group | U-SEMS Group | C-SEMS Group
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 374 days
Description: Definition of adverse event and/or serious adverse event did not differ from the clinicaltrials.gov definitions. All-Cause Mortality - 5 of the 6 participants were followed until their death. Deaths were not related to the study.
Arm/Group | U-SEMS Group | C-SEMS Group
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
Only 6 participants were randomized. A sample size of 96 patients (48 per treatment arm) would be required to detect a 20% difference in stent failure rates at 80% power with an alpha level of 0.05. As 6 participants falls very short of our required sample size, originally planned analysis was not completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT01905384/Prot_SAP_000.pdf